CLINICAL TRIAL: NCT04400864
Title: Mediterranean Diet Versus Paleolithic Diet for the Treatment of Non Alcohlic Fatty
Brief Title: Mediterranean Diet Versus Paleolithic Diet for the Treatment of Non Alcohlic Fatty Liver Disease
Acronym: PALMED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, AMIR SHLOMAI, Head of internal medicine department, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0122-19-rmc
Record Dates: First submitted 2020-05-20; First posted 2020-05-26 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean Diet (Experimental): Nutritional guidelines based on the principals of the Mediterranean Diet
  Interventions: Other: Dietary intervention
- Paleolithic Diet (Experimental): Nutritional guidelines based on the principals of thePaleolithic Diet
  Interventions: Other: Dietary intervention

INTERVENTIONS:
Other: Dietary intervention — dietary counseling based on the principals pf the dietary intervention group.

SUMMARY:
Non- alcoholic fatty liver disease (NAFLD) is one of metabolic syndrome manifestation, and has become the leading cause for cirrhosis and the need for liver transplantation.

The Mediterranean diet showed in many trials its benefit in the treatment of the metabolic syndrome and NAFLD. The Paleolithic Diet includes meat, fish, fruits, vegetables, nuts and seeds and avoidance of processed food and most of carbohydrates. In some studies this diet seemed to decrease triglycerides levels and improve insulin resistance.

The aim of this study is to evaluate the influance of the paleolithic diat for the treatment of NAFLD, as shown in the Mediterranean Diet.

DETAILED DESCRIPTION:
Recruitment of 60 patients with the diagnosis NAFLD from clinics in Rabin Medical center, aged 18-65.

Two study groups- Mediterranean Diet and Paleolithic Diet The dietitian will assign randomly for the study groups, and will assess diet adherence within 6 weeks of the trial and in its end- after 3 months.

blood test for liver enzymes, lipids, crp, mda and HbA1C, will be taken at recruitment and after 3 months.

Ultrasound and elastography will be tested at recruitment and after 3 months, to evaluate the degree of the fatty liver, by a the same doctor who is blind to the study groups.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD

Exclusion Criteria:

* pregnancy
* Chronic kidney disease
* post transplant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the severity of the fatty liver measured by ultrasound and elastography. | 3 months
  Changes in fatty liver severity score according to ultrasound wave intensity analysis- light ; moderate ; severe.

SECONDARY OUTCOMES:
Changes in HbA1C | 3 months
  Blood tests for HbA1C are taken at the beginning and the end of the trial, and analyzed for changes.
Changes in Triglycerides levels | 3 months
  Blood tests for Triglycerides are taken at the beginning and the end of the trial, and analyzed for changes.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Shlomai, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No